CLINICAL TRIAL: NCT06788613
Title: Beyond-FRONTIER: Utilising Hull Lung Health Study Data to Investigate the Performance of TidalSense Diagnostic Algorithms to Identify COPD and Pre-COPD Among Participants in the FRONTIER Programme
Brief Title: Utilising Hull Lung Health Study Data to Investigate the Performance of TidalSense Diagnostic Algorithms to Identify COPD and Pre-COPD Among Participants in the FRONTIER Programme.
Status: Not yet recruiting | Type: Observational
Sponsor: Chiesi UK (Industry)
Collaborators: Hull University Teaching Hospitals NHS Trust (Other Government); TidalSense (Industry); Asthma + Lung UK (Unknown)
Responsible Party: Sponsor
Other Study IDs: Beyond-FRONTIER
Record Dates: First submitted 2024-09-18; First posted 2025-01-23 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-01

CONDITIONS: COPD; Emphysema or COPD; Emphysema
Keywords: COPD; Hull Lung Health; TidalSense; N-tidal
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood biomarker profiles (obtained from the Hull Lung Health Study data) of people with i) confirmed COPD, ii) pre-COPD, and iii) no evidence of COPD will be investigated to explore a potential role for blood biomarkers in COPD diagnostics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Head-to-head comparison with post-bronchodilator spirometry among FRONTIER programme participants: 1. To assess the performance of TidalSense COPD Diagnostic Algorithms for COPD diagnosis in a real-world, head-to-head comparison with post-bronchodilator spirometry among FRONTIER programme participants.
  2. To assess the performance of TidalSense COPD Diagnostic Algorithms for identification of pre-COPD.
  3. Evaluate TidalSense COPD Diagnostic Algorithms ability to identify those at risk of developing COPD within 1-year.
- Explore the blood biomarker profile among FRONTIER study participants to explore COPD identification: 1. Investigate the blood biomarker profile (obtained from the Hull Lung Health Study data) of people with i) confirmed COPD, ii) pre-COPD, and iii) no evidence of COPD.
  2. Explore a potential role for blood biomarkers in COPD diagnostics.

SUMMARY:
Aim: To investigate the potential for N-Tidal to improve COPD diagnosis and enable detection of pre-COPD*.

Objectives:

1. To assess the performance of TidalSense COPD Diagnostic Algorithms for COPD diagnosis in a real-world, head-to-head comparison with post-bronchodilator spirometry among FRONTIER programme participants.
2. To assess the performance of TidalSense COPD Diagnostic Algorithms for identification of pre-COPD.
3. Evaluate TidalSense COPD Diagnostic Algorithms ability to identify those at risk of developing COPD within 1-year.

Aim: Explore the blood biomarker profile among FRONTIER Programme participants to explore a potential role in early COPD identification.

Objectives:

1. Investigate the blood biomarker profile (obtained from the Hull Lung Health Study data) of people with i) confirmed COPD, ii) pre-COPD, and iii) no evidence of COPD.
2. Explore a potential role for blood biomarkers in COPD diagnostics.

   * Pre-COPD is defined, as per the GOLD Report 2023, as individuals who have respiratory symptoms and/or other detectable structural and/or functional abnormalities in the absence of airflow obstruction on forced spirometry. For the purpose of this study, respiratory symptoms will be classified as a CAT score > 10 during FRONTIER clinic attendance and presence of emphysema on low-dose CT considered evidence of structural lung abnormalities

ELIGIBILITY:
All Hull Lung Health Study participants that attend a one-stop diagnostic clinic appointment as part of the FRONTIER Programme (NHS Lung Health Check) will be eligible for inclusion in this study.

Prospective consent provided for use of data for research purposes and for future contact as part of the Hull Lung Health Study

Inclusion criteria:

* Participants in the Hull Lung Health Check Programme (ever smokers aged 55-75 and registered with a Hull GP) with one or more of the following symptoms during their lung health check:
* Breathlessness
* Cough
* Bronchitis
* Recurrent infections
* AND/OR evidence of Emphysema on Low Dose CT

Exclusion criteria:

-Existing COPD diagnosis noted at the time of their Lung Health Check or new COPD diagnosis since Lung Health Check attendance AND prescribed appropriate COPD therapy.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hull Lung Health Study participants that take part in the FRONTIER Programme will be included in this study.
  The FRONTIER Programme is a Collaborative Working Project between the NHS (Hull University Teaching Hospitals NHS Trust) and Chiesi LTD. It aims to enable early COPD diagnosis and timely initiation of evidence-based pharmacological and non-pharmacological interventions to improve outcomes for participants of the Hull Lung Health Check Programme, and the linked Hull Lung Health Study, that missed out on spirometry during their initial Lung Health Check due to infection control precautions
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
To assess the performance of TidalSense COPD Diagnostic Algorithms for COPD diagnosis in a real-world, head-to-head comparison with post-bronchodilator spirometry among FRONTIER programme (NHS Lung Health Check) participants. | 1 year
  We will investigate the performance of TidalSense COPD Diagnostic Algorithms (including the sensitivity, specificity, positive predictive value and negative predictive value of TidalSense 'likely' or 'highly likely' outputs) for COPD diagnosis in a real-world, head-to-head comparison with post-bronchodilator spirometry among NHS Lung Health Check participants. It is anticipated that ~900 patients will participate in the programme.
To assess the performance of TidalSense COPD Diagnostic Algorithms for identification of pre-COPD. | 1 year
  We will investigate the sensitivity, specificity, positive predictive value and negative predictive value of TidalSense 'likely' or 'highly likely' outputs for identifying those that go onto receive a diagnosis of COPD within 1-year of initial review (Pre COPD).
Evaluate TidalSense COPD Diagnostic Algorithms ability to identify those at risk of developing COPD within 1-year | 1 year
  We will investigate the sensitivity, specificity, positive predictive value and negative predictive value of TidalSense 'likely' or 'highly likely' outputs for identifying those at risk of developing COPD within 1-year

SECONDARY OUTCOMES:
Explore a potential role for blood biomarkers in COPD diagnostics including investigating the blood biomarker profile (obtained from the Hull Lung Health Study data) of people with i) confirmed COPD, ii) pre-COPD, and iii) no evidence of COPD | 1 year
  blood biomarker profiles (eosinophils, nTProBNP, fibrinogen, CRP, and IL-6) will be reported descriptively for those with confirmed COPD, pre-COPD and no COPD. Initial univariable pre-screening will inform variable inclusion in a multivariable logistic regression model to explore factors associated with COPD and pre-COPD diagnosis. Identified associated factors will be considered for inclusion in Tidalsense's diagnostic algorithms and the impact on performance investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Micheal Crooks, Prof, Principal Investigator — Hull York Medical School; Karen Watkins, Study Chair — Hull University Teaching Hospitals NHS Trust

IPD SHARING:
Plan to Share IPD: No
Clinical and COPD status data will be retained within the Hull Lung Health Study dataset (held by Hull University Teaching Hospitals NHS Trust) prior to pseudonymisation and transfer to the University of Hull Data Safe Haven. N-Tidal data will be pseudonymised at the point of collection and transferred to the TidalSense cloud where it will be analysed and held by TidalSense. Hull Lung Health Study Data will be available for external research purposes via application to the research team.